CLINICAL TRIAL: NCT01161238
Title: Measuring and Controlling In-Socket Residual Limb Volume Fluctuation
Brief Title: Amputee Residual Limb Volume Fluctuation
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joan Sanders, Professor, University of Washington
Other Study IDs: 30863-E/B; R01HD060585 (NIH)
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower-limb amputee: Subjects with at least one lower limb amputated at the trans-tibial level
  Interventions: Other: Monitored for limb volume

INTERVENTIONS:
Other: Monitored for limb volume — Subjects are monitored for limb volume change using bioimpedance analysis

SUMMARY:
The goal of this project is a useful clinical instrument for diagnosis and treatment of residual limb volume fluctuation in individuals who use prosthetic limbs. One hypothesis to be tested is that the instrument effectively measures short and long term volume fluctuations in individuals with trans-tibial amputation. Another hypothesis to be tested is that when subjects add a sock or insert to the prosthesis residual limb volume decreases, and when they remove the sock or insert residual limb volume increases.

ELIGIBILITY:
Inclusion Criteria:

* trans-tibial amputees who have a regular prosthetist and who wear the prosthesis at least five hours per day.

Exclusion Criteria:

* Inability to ambulate continuously with a prosthesis (with or without the use of an assistive device such as a cane or walker) for 10 minutes indoors on a level walkway. 2. Inability to shift from horizontal to vertical posture in 30 seconds.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people with lower limb amputation that are ambulatory
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Residual limb fluid volume | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Bioengineering Department, Seattle, Washington, United States

REFERENCES:
- [Background] Sanders JE, Harrison DS, Allyn KJ, Myers TR. Clinical utility of in-socket residual limb volume change measurement: case study results. Prosthet Orthot Int. 2009 Dec;33(4):378-90. doi: 10.3109/03093640903214067. PMID 19961297